CLINICAL TRIAL: NCT03892772
Title: Combination Pharmacological Interventions for Multiple Mechanisms of Obstructive Sleep Apnea
Acronym: ComboPlus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Apnimed (Industry)
Responsible Party: Principal Investigator, Scott Aaron Sands, Assistant Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019P000421
Record Dates: First submitted 2019-03-26; First posted 2019-03-27 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- SAS0421a, SAS0421b and SAS0421c (Experimental): Participants will take SAS0421a, SAS0421b and SAS0421c for 3 days. Half doses will be given on the first night.
  Interventions: Drug: SAS0421a; Drug: SAS0421b; Drug: SAS0421c
- SAS0421a and SAS0421b (Active Comparator): Participants will take SAS0421a and SAS0421b for 3 days. Half doses will be given on the first night.
  Interventions: Drug: SAS0421a; Drug: SAS0421b
- SAS0421c (Active Comparator): Participants will take SAS0421c for 3 days. Half doses will be given on the first night.
  Interventions: Drug: SAS0421c
- Placebo (Placebo Comparator): Participants will take placebos for 3 days.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: SAS0421a — treatment will be given for 3 days
  Arms: SAS0421a and SAS0421b; SAS0421a, SAS0421b and SAS0421c
Drug: SAS0421b — treatment will be given for 3 days
  Arms: SAS0421a and SAS0421b; SAS0421a, SAS0421b and SAS0421c
Drug: SAS0421c — treatment will be given for 3 days
  Arms: SAS0421a, SAS0421b and SAS0421c; SAS0421c
Drug: placebo — placebo will be given for 3 days
  Arms: Placebo

SUMMARY:
Currently, there is no pharmacological intervention for OSA that targets multiple pathophysiological deficits in combination. Here the investigators study the effect on sleep apnea severity of combinations of pharmacological agents that stimulate the pharyngeal muscles, stabilize ventilatory control, and increase the arousal threshold.

DETAILED DESCRIPTION:
The primary goal of the current study is to determine the effect of combination therapy targeting phenotypic traits on OSA severity. Specifically, the investigators will assess the effect of combination pharmacological therapy on OSA severity as measured by the apnea-hypopnea index and the arousal index (co-primary outcome variables).

The investigators will also estimate the effects of the interventions on the physiological traits responsible for OSA using polysomnography, namely:

* Pharyngeal anatomy and its propensity towards collapse
* The ability of the upper airway dilator muscles to activate and reopen the airway during sleep (i.e. neuromuscular compensation)
* Arousal threshold from sleep (i.e. the propensity for hypopneas/apneas to lead to arousal and fragmented sleep).
* Stability of the ventilatory control system feedback loop (i.e. loop gain). Baseline traits will be used to examine whether patient characteristics influence the responses to each combination of interventions (i.e. muscles, muscles plus loop gain, muscles plus arousal threshold).

ELIGIBILITY:
Inclusion criteria:

* Ages 18 - 79 years
* Suspected or diagnosed OSA

Exclusion criteria:

* Any uncontrolled medical condition
* Current use of the medications under investigation
* Use of medications expected to stimulate or depress respiration (including opioids, barbiturates, doxapram, almitrine, theophylline, 4-hydroxybutanoic acid).
* Current use of hypnotic medications (trazodone, eszopiclone, benzodiazepines).
* Current use of SNRIs/SSRIs or anticholinergic medications.
* Conditions likely to affect obstructive sleep apnea physiology: neuromuscular disease or other major neurological disorder, heart failure (also below), or any other unstable major medical condition.
* Respiratory disorders other than sleep disordered breathing:

chronic hypoventilation/hypoxemia (awake SaO2 < 92% by oximetry) due to chronic obstructive pulmonary disease or other respiratory conditions.

* Other sleep disorders: periodic limb movements (periodic limb movement arousal index > 10/hr), narcolepsy, or parasomnias.
* Contraindications for SAS0421a and SAS0421b, including:

  * hypersensitivity to SAS0421a and SAS0421b (angioedema or urticaria)
  * pheochromocytoma
  * use of monoamine oxidase inhibitors
  * benign prostatic hypertrophy, urinary retention
  * untreated narrow angle glaucoma
  * bipolar disorder, mania, psychosis
  * history of major depressive disorder (age<24).
  * history of attempted suicide or suicidal ideation within one year prior to screening
  * clinically significant constipation, gastric retention
  * pre-existing seizure disorders
  * clinically-significant kidney disorders (eGFR<60 ml/min/1.73m2)
  * clinically-significant liver disorders
  * clinically-significant cardiovascular conditions
  * severe hypertension (SBP>180 mmHg or DBP>110 mmHg measured at baseline)
  * cardiomyopathy (LVEF<50%) or heart failure
  * advanced atherosclerosis
  * history of cerebrovascular events
  * history of cardiac arrhythmias e.g., atrial fibrillation, QT prolongation
  * other serious cardiac conditions that would raise the consequences of an increase in blood pressure or heart rate
  * myasthenia gravis
  * pregnancy/breast-feeding
* Additional contraindications for SAS0421c, including:

  * Use more than 500 mg/day of Aspirin
  * Allergies to this drug class
  * Adrenocortical insufficiency
  * Low sodium or potassium
  * hyperchloremic acidosis
* Claustrophobia
* Pregnancy or nursing

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2021-07-03 (Actual); Study Completion 2021-07-03 (Actual)

PRIMARY OUTCOMES:
Apnea-hypopnea index [AHI] | 3 days
  Apneas and hypopneas per hour (3% desat and/or arousal), % change from baseline

SECONDARY OUTCOMES:
Hypoxic Burden | 3 days
  Desaturation area under curve × event frequency
Arousal Index | 3 days
  Number of arousals per hour (>=3-sec), % change from baseline
Visual Analog Scale for Sleep Quality | 3 days
  Sleep Quality 0-10 scale, 0 worst sleep quality, 10 best sleep quality
Visual Analog Scale for Waking Unrefreshed | 3 days
  Waking Unrefreshed 0-10 scale, 0 extremely refreshed, 10 extremely unrefreshed

OTHER OUTCOMES:
Visual Analog Scale for Excessive Fatigue | 3 days
  Excessive Fatigue 0-10 scale, 0 no fatigue, 10 highly fatigued
Visual Analog Scale for Low Energy | 3 days
  Low Energy 0-10 scale, 0 no trouble with energy, 10 extremely low energy
Visual Analog Scale for Treatment Satisfaction | 3 days
  Treatment Satisfaction 0-10 scale, 0 extremely dissatisfied, 10 extremely satisfied
Proportion of Total Sleep Time in non-REM Stage 1 | 3 days
  % Total sleep time

CONTACTS AND LOCATIONS:
Overall Officials: Scott A Sands, PhD, Principal Investigator — Brigham and Women's Hospital; Bradley A Edwards, PhD, Principal Investigator — Monash University
Locations (2):
- Brigham and Women's Hospital, Boston, Massachusetts, United States
- Monash University, Clayton, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
Will IPD be available? Yes What data will be shared? All IPD collected during the study, after deidentification.
  When will data be available? Immediately after publication. No end date. With whom? Researchers who provide a methodologically sound proposal. For what types of analyses? Any purpose.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Immediately after publication. No end date.
Access Criteria: 1-page proposals should be directed to Dr. Scott Sands (sasands@bwh.harvard.edu). To gain access, requestors will be asked to sign a data use agreement.

REFERENCES:
- [Derived] Hynes DJ, Mann DL, Landry SA, Joosten SA, Edwards BA, Hamilton GS. Night-to-night variability in obstructive sleep apnea severity, the physiological endotypes, and the frequency of flow limitation. Sleep. 2025 Apr 11;48(4):zsae295. doi: 10.1093/sleep/zsae295. PMID 39688178
- [Derived] Sands SA, Collet J, Gell LK, Calianese N, Hess LB, Vena D, Azarbarzin A, Bertisch SM, Landry S, Thomson L, Joosten SA, Hamilton GS, Edwards BA. Combination pharmacological therapy targeting multiple mechanisms of sleep apnoea: a randomised controlled cross-over trial. Thorax. 2024 Feb 15;79(3):259-268. doi: 10.1136/thorax-2023-220184. PMID 38286618